CLINICAL TRIAL: NCT06326268
Title: Validation of the Improvement in the Management of Chemo-induced Mucositis in Hematology Through the Contribution of Photobiomodulation - The PHOTO-TREAT Study
Brief Title: Interest of Light Therapy in Hematology - The PHOTO-TREAT Study
Acronym: PHOTO-TREAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de cancérologie Strasbourg Europe (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-019; 2023-A02133-42 (Other: ID-RCB Number)
Record Dates: First submitted 2024-03-11; First posted 2024-03-22 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Leukemia, Myeloid, Acute; Lymphoma
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Photobiomodulation (Other): • Patients: In induction of acute myeloblastic leukemia OR Allografts in first remission with myeloablative conditioning OR Autografts in the context of aggressive lymphoma;
  Interventions: Device: Phototherapy system CareMin650TM

INTERVENTIONS:
Device: Phototherapy system CareMin650TM — * As part of preventive treatment: Photobiomodulation sessions will be carried out at a dose of 3 joules for 1 minute 51 seconds, 3 times a week (for a maximum duration of 4 to 6 weeks).
  * As part of curative treatment (i.e. for patients developing mucositis, from grade I): photobiomodulation will be carried out at a curative dose of 6 joules daily (for a maximum duration of 4 to 6 weeks ) for 3 minutes 34 seconds.

SUMMARY:
Chemo-induced mucositis is a common complication in patients treated for hematologic malignancies. They can manifest itself as a simple local irritation with erythema and inflammation but can also progress to erosions and ulcerations of the entire oral mucosa and are also responsible for an increased risk of infection in these immunocompromised patients.

The only therapies currently offered are local care and intravenous analgesics. Studies in pediatric hematology show the effectiveness of prevention and low-dose laser treatment in chemo-induced mucositis, both in terms of reducing the number of mucositis developed but also in terms of reducing the grade of mucositis. This currently results in a recommendation for the use of photobiomodulation by international bodies such as ESMO (European Society for Medical Oncology).

DETAILED DESCRIPTION:
During this research, the investigators aim at validating the efficacy and impact of photo-biomodulation in the management of chemo-induced mucositis in hematology department of Strasbourg Cancer Institute (ICANS).

ELIGIBILITY:
Inclusion Criteria:

* Adult patient;
* Patients:

In induction of acute myeloblastic leukemia OR Allografts in first remission with myeloablative conditioning OR Autografts in the context of aggressive lymphoma;

* Signature of informed consent;
* Patient registered with social security.

Exclusion Criteria:

* Patient under guardianship or curatorship
* Pregnant and breastfeeding woman
* Allergy to polyurethanes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2025-09-17 (Estimated); Study Completion 2025-09-17 (Estimated)

PRIMARY OUTCOMES:
Evaluate the impact of Photobiomodulation (PBM) therapy in the management of chemo-induced mucositis in terms of prevalence of mucositis | Up to 12 weeks
  Rate of occurrence of mucositis, graded according to NCI-CTCAE V5.0 criteria

SECONDARY OUTCOMES:
Evaluate the impact of PBM in the management of chemo-induced mucositis in terms of reduction in analgesic consumption. | Up to 12 weeks
  Consumption of level III analgesics during aplasia after chemotherapy.
Evaluate the impact of PBM in terms of infection by bacterial translocation risk reduction. | Up to 12 weeks
  Consumption of systemic anti-infectives during aplasia after induction and conditioning chemotherapy.
Evaluate the impact of PBM in terms of reduction of the use of artificial feeding. | Up to 12 weeks
  Duration of artificial nutrition during aplasia
Evaluate the impact of PBM in terms of reduction of the length of hospital stay. | Up to 12 weeks
  Length of hospitalization
Evaluate the impact of PBM in terms of reduction of the number of transfusions. | Up to 12 weeks
  Number of transfusions during hospitalization
Evaluate the impact of PBM in terms of pain reduction | Up to 12 weeks
  Assessment using a visual analogue scale (VAS, graded from 0 to 10). Measurement before and after each PBM session.
Evaluate the impact of PBM on patient's satisfaction regarding pain management during hospital stay | Up to 12 weeks
  Evaluation of patient satisfaction with the hospital stay - questions on pain management from the Picker Patient Experience Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Anne ZILLIOX, MD, Principal Investigator — Institut de cancérologie Strasbourg Europe
Locations (1):
- Institut de cancérologie Strasbourg Europe, Strasbourg, France

REFERENCES:
- [Background] Buclin CP, Uribe A, Daverio JE, Iseli A, Siebert JN, Haller G, Cullati S, Courvoisier DS. Validation of French versions of the 15-item picker patient experience questionnaire for adults, teenagers, and children inpatients. Front Public Health. 2024 Feb 19;12:1297769. doi: 10.3389/fpubh.2024.1297769. eCollection 2024. PMID 38439757